CLINICAL TRIAL: NCT07357558
Title: A Qualitative Study Investigating the Lived Experiences and Impact of Reproductive Issues in Adults With Primary Ciliary Dyskinesia
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM O&G0332
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Primary Ciliary Dyskinesia (PCD)
Keywords: fertility; pregnancy; reproduction; parenthood; qualitative; interviews
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview only — No intervention

SUMMARY:
Study involving undertaking research interviews with adults who have primary ciliary dyskinesia in the UK about their views and experiences of fertility, pregnancy and parenthood

ELIGIBILITY:
Inclusion Criteria:

* Lives in United Kingdom
* 'likely' or 'confirmed' diagnosis of PCD
* able and willing to sign the consent form

Exclusion Criteria:

* unwilling to participate in the study
* not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with primary ciliary dyskinesia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative description of views and experiences of participants | Explored during study interview (day 1)
  Explored during study interview

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Southampton NHS Trust, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided